CLINICAL TRIAL: NCT02186457
Title: Routine Antibiotic Irrigation in Patients Undergoing Pancreatoduodenectomy to Reduce Infection and Fistula Rates
Brief Title: Antibiotic Irrigation for Pancreatoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael G. House, Associate Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1403644165
Record Dates: First submitted 2014-07-01; First posted 2014-07-10 (Estimated); Results first posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: Surgery; Infection
Keywords: Pancreatoduodenectomy; Whipple
MeSH Terms: conditions — Infections | interventions — Polymyxin B; Saline Solution; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polymyxin B in Normal Saline (Experimental): Polymyxin B (500,000 U) in 1 liter of 0.9% Normal Saline
  Interventions: Drug: Polymyxin B in Normal Saline
- Placebo: Normal Saline (Placebo Comparator): 0.9 % Normal Saline
  Interventions: Other: Placebo: Normal Saline

INTERVENTIONS:
Drug: Polymyxin B in Normal Saline — Antibiotic irrigation via peritoneal lavage
  Other Names: Antibiotic
  Arms: Polymyxin B in Normal Saline
Other: Placebo: Normal Saline — Placebo irrigation via peritoneal lavage
  Other Names: Placebo
  Arms: Placebo: Normal Saline

SUMMARY:
The purpose of this study is to determine if the routine use of antibiotic irrigation during pancreas surgery (Whipple procedure) will decrease superficial and organ space infections.

DETAILED DESCRIPTION:
The primary aim of this study is to test the efficacy of routine antibiotic irrigation in reducing superficial and organ space infections among patients undergoing pancreatoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and older;
* Open pancreatoduodenectomy for any diagnosis

Exclusion Criteria:

* Pregnant;
* Prisoners;
* Patients undergoing concomitant colectomy;
* Antibiotic allergy to study medication;
* Serum creatinine > 2.0;
* Unable to provide informed consent

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael House, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: more patients enrolled
Period: Overall Study
Arm/Group | Polymyxin B in Normal Saline | Placebo: Normal Saline
Started | 95 | 95
Completed | 95 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polymyxin B in Normal Saline | Placebo: Normal Saline | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Categorical [Count of Participants; unit: Participants]
  Age distribution: <=18 years | 0 | 0 | 0
  Age distribution: Between 18 and 65 years | 60 | 55 | 115
  Age distribution: >=65 years | 35 | 40 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (1.3) | 64.4 (1.5) | 64.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 55 | 57 | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 90 | 88 | 178
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 95 | 95 | 190

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Infections
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Polymyxin B in Normal Saline | Placebo: Normal Saline
Number analyzed (Participants) | 95 | 95
Participants | 11 | 10

2. Secondary Outcome: The Number of Patients With Fistulas
Time Frame: 5 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Polymyxin B in Normal Saline | Placebo: Normal Saline
Number analyzed (Participants) | 95 | 95
Participants | 25 | 29

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Polymyxin B in Normal Saline | Placebo: Normal Saline
All-Cause Mortality (participants affected / at risk) | 1/95 | 2/95
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/95
Other Adverse Events (participants affected / at risk) | 0/95 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT02186457/Prot_SAP_000.pdf